CLINICAL TRIAL: NCT03285100
Title: Pilot Study to Assess the Effects of Discontinuation of Vitamin K Antagonists on the Rate of Elastin Degradation
Brief Title: The Effects of Discontinuation of Vitamin K Antagonists on the Rate of Elastin Degradation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Canisius-Wilhelmina Hospital (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Rob Janssen, MD, PhD, Canisius-Wilhelmina Hospital
Other Study IDs: NL60536.091.17
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Emphysema or COPD; Aneurysm; Cystic Fibrosis; Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Aneurysm; Cystic Fibrosis; alpha 1-Antitrypsin Deficiency | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * at baseline: blood sample of 15mL (EDTA-plasma), divided in four two portions (one for determination of dp-ucMGP and one for desmosine)
  * at baseline: blood sample of 10mL (EDTA-plasma). DNA will be isolated from these samples for determination of the VKORC1 polymorphisms
  * after six months: blood sample of 15mL (EDTA-plasma), divided in four two portions (one for determination of dp-ucMGP and one for desmosine)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Venipuncture — * Approximately 6 months after discontinuation of VKAs one additional venipuncture will be performed for determination of dp-ucMGP and desmosine.
  * At baseline two additional blood collection tubes will be drawn for determination of dp-ucMGP, desmosine and VKORC1 polymorphisms. Since this is during one of the last regular International Normalized Ratio (INR) testing at the anticoagulation clinic, no additional venipuncture has to be performed at this moment.

SUMMARY:
Background: Elastin is a unique protein providing elasticity, resilience and deformability to dynamic tissues, such as lungs and vasculature. Elastin fibers are characterized by their high affinity for calcium. However, calcified elastin is more prone to the degrading effects of proteases and, in turn, partially degraded elastin has an even higher affinity for calcium. A disturbed balance between proteases and anti-proteases is a major underlying mechanism in the development of chronic obstructive pulmonary disease (COPD). Virtually the only protein that can protect elastin from calcification is matrix Gla-protein (MGP), which needs vitamin K for its activation. In COPD patients, a lower vitamin K status is found when compared to control subjects and an inverse association exists between vitamin K status and elastin degradation. In addition, vitamin K status is lower and elastin degradation is accelerated in Vitamin K antagonist (VKA) users.

VKAs are widely used. Nowadays, an increasing number of patients uses direct oral anticoagulants (DOACs), which do not influence vitamin K status. The hypothesis of this study is that discontinuation of VKAs results in an improved vitamin K status and deceleration of elastin degradation. In order to test this hypothesis, an observational pilot study will be conducted in which the change in elastin degradation- quantified by plasma desmosine concentrations - in patients who discontinue use of VKAs will be used as primary endpoint.

Study design: Observational study. Study population: A total of 30 VKA users who will discontinue the use of VKAs. Elastin degradation rate (quantified by plasma desmosine levels) and vitamin K status (quantified by measuring plasma levels of dephosphorylated uncarboxylated (dp-uc)MGP) will be measured during the use of VKAs and approximately 6 months after discontinuation of VKAs. Furthermore, the VKORC1 polymorphisms will be determined.

Main study parameters: The primary endpoint is the change in the rate of elastin degradation quantified by the plasma desmosine assay. Secondary endpoints are the change in vitamin K status quantified by measuring plasma levels of dp-ucMGP, the relation between desmosine and dp-ucMGP and differences of desmosine and dp-ucMGP levels among subjects with different polymorphisms of the vitamin K 2,3-epoxide reductase complex 1 (VKORC1) gene.

ELIGIBILITY:
Inclusion Criteria:

* Use of VKAs for at least 3 months
* Stop VKAs at short time
* Written informed consent
* Age ≥18 years
* Ability to comply with all study requirements

Exclusion Criteria:

* Active malignancy or cured malignancy <12 months prior to enrollment
* Use of maintenance dose oral corticosteroids
* Serious mental impairment
* Life expectation of less than 6 months on the basis of concurrent disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 VKA users from the anticoagulant clinic in the Canisius Wilhelmina Hospital, who are going to discontinue the use of VKAs at short time
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference in elastin degradation rate | Plasma desmosine is measured at baseline and 6 months after discontinuation of VKAs
  Difference in elastin degradation rate before and after discontinuation of VKAs, quantified by the change in plasma desmosine levels

SECONDARY OUTCOMES:
Difference in vitamin K status | Plasma dp-ucMGP is measured at baseline and 6 months after discontinuation of VKAs
  Difference in vitamin K status before and after discontinuation of VKAs, quantified by the change in dp-ucMGP, discontinuation of VKAs.
Association between desmosine and dp-ucMGP | Desmosine and dp-ucMGP are determined before discontinuation of VKAs and 6 months after discontinuation of VKAs
  Association between desmosine and dp-ucMGP both in patients who use VKAs and do not use VKAs.
Differences in desmosine and dp-ucMGP levels between different VKORC1 polymorphisms | Desmosine and dp-ucMGP are determined, both before discontinuation of VKAs and 6 months after discontinuation of VKAs. VKORC1 polymorphisms are determined before discontinuation of VKAs.
  Levels of dp-ucMGP and desmosine levels of subjects with different VKORC1 polymorphisms are compared, both during the use of VKAs and after discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Janssen, MD, PhD, Principal Investigator — Canisius-Wilhelmina Hospital
Locations (1):
- Canisius Wilhelmina Hospital, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mithieux SM, Weiss AS. Elastin. Adv Protein Chem. 2005;70:437-61. doi: 10.1016/S0065-3233(05)70013-9. PMID 15837523
- [Background] Robert L, Robert AM, Fulop T. Rapid increase in human life expectancy: will it soon be limited by the aging of elastin? Biogerontology. 2008 Apr;9(2):119-33. doi: 10.1007/s10522-007-9122-6. Epub 2008 Jan 4. PMID 18175202
- [Background] Bouvet C, Moreau S, Blanchette J, de Blois D, Moreau P. Sequential activation of matrix metalloproteinase 9 and transforming growth factor beta in arterial elastocalcinosis. Arterioscler Thromb Vasc Biol. 2008 May;28(5):856-62. doi: 10.1161/ATVBAHA.107.153056. Epub 2008 Feb 21. PMID 18292396
- [Background] Basalyga DM, Simionescu DT, Xiong W, Baxter BT, Starcher BC, Vyavahare NR. Elastin degradation and calcification in an abdominal aorta injury model: role of matrix metalloproteinases. Circulation. 2004 Nov 30;110(22):3480-7. doi: 10.1161/01.CIR.0000148367.08413.E9. Epub 2004 Nov 15. PMID 15545515
- [Background] Turino GM, Ma S, Lin YY, Cantor JO, Luisetti M. Matrix elastin: a promising biomarker for chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2011 Sep 15;184(6):637-41. doi: 10.1164/rccm.201103-0450PP. PMID 21757624
- [Background] Maclay JD, McAllister DA, Rabinovich R, Haq I, Maxwell S, Hartland S, Connell M, Murchison JT, van Beek EJ, Gray RD, Mills NL, Macnee W. Systemic elastin degradation in chronic obstructive pulmonary disease. Thorax. 2012 Jul;67(7):606-12. doi: 10.1136/thoraxjnl-2011-200949. Epub 2012 Feb 28. PMID 22374923
- [Background] Williams MC, Murchison JT, Edwards LD, Agusti A, Bakke P, Calverley PM, Celli B, Coxson HO, Crim C, Lomas DA, Miller BE, Rennard S, Silverman EK, Tal-Singer R, Vestbo J, Wouters E, Yates JC, van Beek EJ, Newby DE, MacNee W; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) investigators. Coronary artery calcification is increased in patients with COPD and associated with increased morbidity and mortality. Thorax. 2014 Aug;69(8):718-23. doi: 10.1136/thoraxjnl-2012-203151. Epub 2014 Jan 28. PMID 24473329
- [Background] Geleijnse JM, Vermeer C, Grobbee DE, Schurgers LJ, Knapen MH, van der Meer IM, Hofman A, Witteman JC. Dietary intake of menaquinone is associated with a reduced risk of coronary heart disease: the Rotterdam Study. J Nutr. 2004 Nov;134(11):3100-5. doi: 10.1093/jn/134.11.3100. PMID 15514282
- [Background] Knapen MH, Braam LA, Drummen NE, Bekers O, Hoeks AP, Vermeer C. Menaquinone-7 supplementation improves arterial stiffness in healthy postmenopausal women. A double-blind randomised clinical trial. Thromb Haemost. 2015 May;113(5):1135-44. doi: 10.1160/TH14-08-0675. Epub 2015 Feb 19. PMID 25694037
- [Background] Patillon B, Luisi P, Blanche H, Patin E, Cann HM, Genin E, Sabbagh A. Positive selection in the chromosome 16 VKORC1 genomic region has contributed to the variability of anticoagulant response in humans. PLoS One. 2012;7(12):e53049. doi: 10.1371/journal.pone.0053049. Epub 2012 Dec 28. PMID 23285254
- [Background] Rabinovich RA, Miller BE, Wrobel K, Ranjit K, Williams MC, Drost E, Edwards LD, Lomas DA, Rennard SI, Agusti A, Tal-Singer R, Vestbo J, Wouters EF, John M, van Beek EJ, Murchison JT, Bolton CE, MacNee W, Huang JT; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Circulating desmosine levels do not predict emphysema progression but are associated with cardiovascular risk and mortality in COPD. Eur Respir J. 2016 May;47(5):1365-73. doi: 10.1183/13993003.01824-2015. Epub 2016 Mar 23. PMID 27009168

DOCUMENTS (2):
  • Informed Consent Form (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT03285100/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT03285100/Prot_SAP_001.pdf